CLINICAL TRIAL: NCT01330498
Title: Longitudinal Pharmacokinetic, Pharmacodynamic, Immunological, and Biochemical Sample Collection With MRI and Relapse Analysis of a Tysabri Patient Cohort
Brief Title: Longitudinal Pharmacokinetic, Pharmacodynamic, Immunological, and Biochemical
Status: Completed | Type: Observational
Sponsor: John F. Foley, MD (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor-Investigator, John F. Foley, MD, Sponsor-Ivestigator, Rocky Mountain MS Research Group, LLC
Organization: Rocky Mountain MS Research Group, LLC (Other)
Other Study IDs: 001-002-TY
Record Dates: First submitted 2011-03-31; First posted 2011-04-07 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Multiple Sclerosis
Keywords: Longitudinal assessment of biomarkers; duration of natalizumab; stratification of risk for PML
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum for PK/PD, SVCAM back-up samples will be kept.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tysabri (natalizumab) infusing: Patients with relapsing forms of MS who participated in 001-001-TY and are currently still infusing with Tysabri (natalizumab).

SUMMARY:
This is an open-label study of patients with relapsing forms of Multiple Sclerosis designed to assess the longitudinal pharmacokinetic, pharmacodynamic, immunological, and biochemical sample collection with MRI and relapse analysis of a Tysabri patient cohort. The study hopes to identify secondary and tertiary risk stratification markers that would aid in the clinical management of patients who are JC antibody positive.

DETAILED DESCRIPTION:
Progressive multifocal leukoencephalopathy (PML) has been related to the utilization of Tysabri as a therapeutic agent in the treatment of multiple sclerosis. The etiologic agent is the human polyomavirus JC. PML can result from lytic infection of glial cells via a mutant JC virus in multiple sclerosis patients being actively treated with Tysabri. The mutated JC virus is a neurotrophic virus that infects only humans. "The regulatory region sequence of the JC virus is hypervariable and contains determinants for neurotropism and neurovirulence." (Jensen and Major, 2001). In patients initially infected for the most part in childhood the virus tends to remain quiescent in kidneys, bone marrow and lymphoid tissue. The true incidence of JC virus seroprevalance is currently being assessed via two Biogen Idec clinical trials (STRATIFY 1 101JC401 and STRATIFY 2 101JC402). Application has been made to the FDA regarding a label change for Tysabri which will incorporate the use of the JC antibody assay. Upon FDA approval of the label change, the JC assay will serve as a primary risk stratification tool in the clinical use of Tysabri. Secondary and tertiary risk stratification markers would greatly aid in the clinical management of patients who are JC antibody positive.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Aged 18 to 80 years old, inclusive, at the time of informed consent.
* Must be a patient with a relapsing form of Multiple Sclerosis enrolled in the TOUCH Prescribing Program who is not expected to discontinue Tysabri® therapy prior to completion of the requirements of this study.
* Must have participated in IIT I (Foley, IIT 1 001-001-TY) in March, April, or May of 2010.
* Must have a magnetic resonance imaging (MRI) brain scan, performed prior to the initiation of treatment with natalizumab, on file.
* Must weigh between 38 and 180 kg, inclusive.
* Up to 40 patients will be asked to also participate in Part B, the PK/PD subset,
* Approximately fifty patients will be asked to also participate in the sub-study Part C. These patients will have been in the bottom 20th percentile for iATP in Foley IIT 1 001-001-TY.

Exclusion Criteria:

* If subject answers 'Yes" to any question on the PML questionnaire that is not resolved prior to infusion as per standard operating procedure for natalizumab infusion.
* If subject consumes alcohol within 24 hours of blood specimen collection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsing forms of MS. Conducted at one site in the US. Subjects currently enrolled in TOUCH Prescribing Program, and participated in Foley 001-001-TY eligible.
  Subset of approx. 40 patients to participate in Part B. 11 high risk bivalent patients 11 low risk monovalent patients 9 patients who participated in 2009 PK/PD study (Biogen Idec, 101MS406) 9 patients with infusion cycle of 38 days plus or minus 2 days
  Part C "Intracellular energetic in Tysabri therapy":
  Patients whose iATP fell into the bottom 20th percentile will be asked to participate in a sub-study that includes Part A with the addition of collecting iATP. This number is approximately 50 participants.
  Part D patients from 001-001-TY with low or normal IgG4 levels will be asked to participate in sub-study for an additional IgG4 assay collected at 3-5 days post-infusion. This number is approximately 30 participants.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Duration Effect of natalizumab | 18 months
  Primary: To further understand the duration effect of natalizumab at the biochemical, cellular, and pharmacokinetic levels in natalizumab patients; identify biomarkers which could aid in patient risk modification for (PML). Assess the stability of natalizumab concentration via pharmacokinetic measurement in ug/ml.

SECONDARY OUTCOMES:
Stability of cell trafficking inhibition | 18 months
  Secondary endpoint: Assess the stability of cell trafficking inhibition produced through steady state Natalizumab administration through an infusion cycle. Cell trafficking is measured via sVCAM, measurement units ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: John F Foley, MD, Principal Investigator — Rocky Mountain MS Research Group, LLC
Locations (1):
- Rocky Mountain Multiple Sclerosis Clinic, Salt Lake City, Utah, United States